CLINICAL TRIAL: NCT01390298
Title: Pain and Function After Orthopedic Surgery
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00017394
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Chronic Pain
Keywords: chronic pain after knee replacement surgery
MeSH Terms: conditions — Chronic Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Adult patients scheduled for elective unicompartmental or total knee replacement surgery or total hip replacement will be consented to participate
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational study only

SUMMARY:
The purpose of this study is to provide preliminary data for a Program Project Grant to the National Institutes of Health to examine specific explanations regarding identifying patients at risk for chronic pain after surgery and identifying mechanisms which may be altered to decrease this risk.

This study will help investigators better understand chronic pain that develops after surgery. We are proposing to study different factors related to the surgical experience and factors in the environment to determine if any play a role in the development of chronic pain after surgery.

DETAILED DESCRIPTION:
Primary indications for major joint surgery include limited joint function and pain. Although joint replacement or repair surgery is usually remarkably effective, in some cases pain and function are worse or not improved after surgery. Chronic pain after some surgical procedures, e.g., phantom limb pain after extremity amputation, has been long recognized, but more recent investigations suggest that chronic pain after physical injury including that of major surgery is not uncommon. The purpose of this study is to provide preliminary data for a Program Project Grant to the National Institutes of Health to examine specific hypotheses regarding identifying patients at risk for chronic pain after surgery and probing mechanisms which may be manipulated to decrease this risk.

Methods:

Patients who are undergoing elective orthopedic surgery: unicompartmental knee replacement or a total knee replacement will be approached and asked to provide consent to participate in 6 months of observation after their surgery. During this time, participants will not alter their usual treatment in any way (i.e., no treatment algorithms will be altered for this study), but will complete diaries and survey instruments at numerous intervals.

Objectives:

1. To demonstrate the feasibility of conducting this protocol in this clinical population. The execution of this study will allow us to identify expected enrollment rates, patient drop-out rates, and other threats to the accurate assessment of the course of pain after major joint surgery.
2. To estimate the individual variability in pain trajectories over time and to obtain effect size estimates for factors that predict pain trajectory.

Interventions:

The proposed study is a prospective longitudinal observational study. All patients will complete written informed consent.

The following questionnaires will be completed:

Daily Stress Inventory Multidimensional Pain Inventory Catastrophizing Scale of the Coping Strategies Questionnaire Center for Epidemiological Studies Scale of Depression Stait-Trait Anxiety Inventory Pain Anxiety Symptom Scale Pain Medication Attitudes Questionnaire Pain Disability Index Pain Locus of Control Scale Pain Self-Efficacy Scale Marital adjustment test Job Satisfaction Survey Tampa Scale of Kinesiophobia

At Home Diary Assessments Each of the following measures listed below are programmed into an electronic diary (iPod touch) that has been especially programmed for the current study using Pendragon Forms VI.

All participants will complete the assessments in a sequence using one of several methods:

A. Inpatient evaluation (surgery to discharge): Nursing staff will inquire about the patients pain levels using standard of care methods and assessment tools (e.g., numerical rating scale 0 - 10).

B. Ecological Momentary assessment (discharge to day 14): The diary is programmed to emit an alarm at three random times throughout a 12-hour day (i.e., during the patients wake cycle). The patient will then have 10 minutes to complete an entry for that entry to be considered valid (i.e., waiting 2 hours to make an entry is not capturing the random assignment of assessment times).

C. Once daily (day 15 to day 28): The patient is instructed to complete a diary entry at the end of their day, just prior to going to sleep.

D. Once weekly (day 29 to day 85): The patient will be called at their home and participate in a brief interview.

E. Once monthly (day 86 to day 168): The patient will be called at their home and participate in a brief interview once each month.

In addition, information from the postoperative care from the orthopedic surgery division will be recorded, including range of joint motion and functional limitations, if any, at the times of routine postoperative clinic visits. The iPod touch will be returned at the postoperative visit following surgery.

Outcome measures: The primary outcome measure for this study is self-reported pain intensity. To obtain estimates of pain intensity, we will use the McGill Pain Questionnaire - Short Form (MPQ). This instrument has been extensively used to assess pain in a wide variety of settings, and is uniquely suited to our present study in that the items can be completed while in a post-operative setting as well as a daily diary setting.

ELIGIBILITY:
Inclusion Criteria

* American Society of Anesthesiologist (ASA) physical status 1, 2, or 3
* Scheduled for a total knee replacement or unicompartmental knee replacement

Exclusion Criteria:

* ASA >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective unicompartmental, total knee replacement or total hip replacement surgery, will be included. Patients will be American Society of Anesthesiologists physical status 1, 2, or 3.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Adult patients scheduled for elective unicompartmental or total knee replacement surgery or total hip replacment
  Observational: Observational study only
Period: Overall Study
Arm/Group | All Study Participants
Started | 55
Completed | 31
Not Completed | 24
Not completed — Death | 1
Not completed — long term ICU admission | 1
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 7
Not completed — Surgery cancelled | 1

BASELINE CHARACTERISTICS:
Population: Analysis population is based on the 40 participants that were initiated into the study after signing the informed consent.
  55 Consented and 14 withdrew after signing consent and 1 withdrew because surgical procedure canceled leaving a total of 40 participants that completed baseline questionnaires.
Groups:
- All Study Participants: Adult patients scheduled for elective unicompartmental or total knee replacement surgery or total hip replacement will be consented to participate
  Observational: Observational study only
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 60.35 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Pain Intensity
Description: McGill Pain Questionnaire: 0-10 Visual Analog Scale for self reported pain intensity 0= no pain 10= worst pain imaginable Lower score denotes better outcomes
  Visual Analog Scores were obtained during the following times:
  Twice daily: day of hospital discharge through postoperative day 14 Once daily postoperative day 15 through postoperative day 28 Once weekly postoperative day 29 through postoperative day 85 Once monthly postoperative day 86 through postoperative day 168
  Longitudinal analysis of primary outcome measure over time was estimated by longitudinal mixed models and not one mean and standard deviation.
  The change in pain over time was modeled by 7.7344 - 1.6013(log(time))
Time Frame: Day of hospital discharge to postoperative day 168
Population: Lower Extremity Total Joint Arthroplasty (TJS) Cohort (n=31)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
units on a scale | 3 (2.9)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Observational: Adult patients scheduled for elective unicompartmental or total knee replacement surgery or total hip replacment
  Observational: Observational study only
Arm/Group | Observational
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 1/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=31)
Subject experienced myocardial infarction during the immediate postoperative period (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=31)
Subject experienced postoperative complications resulting in long term hospitializaton (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-07-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT01390298/Prot_SAP_000.pdf
  • Informed Consent Form (2013-03-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT01390298/ICF_001.pdf